CLINICAL TRIAL: NCT03717870
Title: Evaluation of Reproductive Outcomes After Different Management of Ovarian Endometrioma Prior to Assisted Reproduction Technology (ART): Laparoscopic Enucleation Vs Prolonged Pituitary Downregulation With Gonadotropin Releasing Hormone (GnRH)-Agonists
Brief Title: Surgery and ART For Endometrioma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFE-1
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Ovarian Endometrioma; Infertility, Female
Keywords: Endometrioma; Infertility; Laparoscopy; GnRH-a; Assisted Reproduction Technology; Reproductive outcomes
MeSH Terms: conditions — Endometriosis; Infertility, Female; Infertility | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Experimental): Laparoscopic enucleation of ovarian endometrioma (stripping of the peripheral capsule and coagulation using the lowest energy source available).
  Interventions: Procedure: Laparoscopic enucleation of ovarian endometrioma.; Procedure: Assisted Reproductive Technology (ART)
- Prolonged pituitary downregulation (Active Comparator): Treatment with GnRH-a (triptorelin, goserelin, and leuprolide), with add-back therapy (combined oral contraceptive) for 3-6 months.
  Interventions: Procedure: Prolonged pituitary downregulation; Procedure: Assisted Reproductive Technology (ART)

INTERVENTIONS:
Procedure: Laparoscopic enucleation of ovarian endometrioma. — Laparoscopic enucleation of ovarian endometrioma (stripping of the peripheral capsule and coagulation using the lowest energy source available).
  Arms: Surgery
Procedure: Prolonged pituitary downregulation — Treatment with GnRH-a (triptorelin, goserelin, and leuprolide), with add-back therapy (combined oral contraceptive) for 3-6 months.
  Arms: Prolonged pituitary downregulation
Procedure: Assisted Reproductive Technology (ART) — Fresh ART cycle: ovarian stimulation, oocyte retrieval, in vitro fertilization and embryo transfer.

SUMMARY:
Endometriosis is an estrogen-dependent chronic disease, characterized by the presence of endometrial-like tissue, glands and stroma outside the uterine cavity. Although endometriosis is classified in four stage (minimal, mild, moderate, severe), from the clinical point of view it is possible to subdivide among peritoneal superficial lesions, ovarian endometriomas and Deep Infiltrating Endometriosis (DIE).

According to the European Society for Human Reproduction and Embryology (ESHRE) Guideline on the management of women with endometriosis, it is recommended to clinicians that in infertile women with endometrioma larger than 3 cm, cystectomy should be considered prior to Assisted Reproduction Technology (ART) to improve endometriosis-associated pain or the accessibility of follicles. They further recommend that clinicians counsel women with endometrioma regarding the risks of reduced ovarian function after surgery, the possible loss of the ovary, and consider that the decision to proceed with surgery should be taken carefully if the woman has had previous ovarian surgery.

In addition, this Guideline suggests that clinicians can prescribe prolonged (3-6 months) pituitary downregulation with Gonadotropin Releasing Hormone-agonists (GnRH-a) prior to ART, in order to increase live birth rate by four-fold.

Despite these recommendations, to date there is not robust evidence to choose between the two strategies prior to ART in order to improve reproductive outcomes.

For this reason, the aim of the current study will be to compare reproductive outcomes in infertile women affected by ovarian endometrioma, undergoing laparoscopic enucleation or prolonged pituitary downregulation with GnRH-a, prior to ART.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ART: compromised tubal function, male factor infertility, other treatments have failed and/or prolonged infertility of more than 4 years.
* Age between 18 and 35 years.
* Ultrasound diagnosis of one ovarian endometriotic cyst with a diameter of 30 mm or more, according to the International Ovarian Tumor Analysis (IOTA)-criteria for reliable diagnosis of endometriomas in premenopausal women.

Exclusion Criteria:

* Any comorbidity other than ovarian endometrioma.
* Deep Infiltrating Endometriosis.
* Previous ovarian surgery.
* Bilateral endometriomas.
* The use of donor oocytes/sperm.
* ART with preimplantation genetic testing, as the number of embryos suitable. for transfer or cryopreservation is significantly lower compared to normal ART.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy with fetal heartbeat | Within 8 weeks from embryo transfer
  Ultrasound-confirmed intrauterine pregnancy with fetal heartbeat

SECONDARY OUTCOMES:
Biochemical pregnancy | Within 8 weeks from embryo transfer
  Positive HCG serum testing
Miscarriage | Within 12 weeks from embryo transfer
  Ultrasound-confirmed abortion
Live birth rate | Within 41 weeks from embryo transfer
  Delivered fetus after 28 gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided